CLINICAL TRIAL: NCT05827900
Title: Metacognitive Training in Individuals at Risk for Psychosis - a Pilot Study
Brief Title: Metacognitive Training in Ultra-high Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nilufar Mossaheb, Assoc.Prof Dr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT in UHR 130323
Record Dates: First submitted 2023-04-11; First posted 2023-04-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ultra-high Risk for Psychosis; Clinical High Risk for Psychosis; At-risk Mental State

STUDY DESIGN:
Intervention Model Description: Randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Metacognitive Group Training
  Interventions: Behavioral: Metacognitive Training
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Metacognitive Training — Minimum of 6 sessions; but planned 10-12 sessions of metacognitive group training
  Arms: Intervention

SUMMARY:
The aim of this pilot study is to examine whether metacognitive training can improve symptoms, wellbeing and functioning in individuals with attenuated psychotic symptoms. Metacognitive group training is an intervention designed to raise awareness on and change cognitive biases that may foster the development of psychotic symptoms such as delusions. It has been shown to be helpful in people with manifest psychosis. The main goal is to assess whether this training is prone to reducing symptoms in individuals at risk for psychosis. Participants will be randomized either to treatment as usual or to treatment as usual plus metacognitive training. Follow-ups will be performed over the period of one year.

DETAILED DESCRIPTION:
Background: Different metacognitive distortions similar to those of patients with schizophrenia could be shown in individuals with attenuated psychotic symptoms at ultra-high risk for psychosis (UHR) including more dysfunctional metacognitive beliefs, overconfidence in judgements, a jumping-to- conclusion reasoning style associated with impaired working memory, a metamemory bias and intolerance of uncertainty. Recent research points towards a positive effect of metacognitive training (MCT) on positive symptoms, data gathering and delusions in patients with schizophrenia by raising awareness for cognitive biases.

Aims: The aim of this study is to examine whether metacognitive training can improve psychopathology in individuals with attenuated psychotic symptoms via changes in metacognitive biases and beliefs. Study design: The study is randomized-controlled, prospective.

Methods: 15 individuals fulfilling UHR criteria will be randomly assigned to a group receiving MCT+treatment as usual (TAU) at an early psychosis clinic for a duration of approximately 8-12 weeks and 15 individuals fulfilling UHR criteria will receive TAU only. Both groups will undergo psychiatric assessments to exclude current or past psychiatric disorders as well as psychosis threshold and current psychopathology. Also, an assessment of IQ, psychosocial functioning and metacognitive biases and beliefs will be done. Assessments will be done at baseline, after 12, 26 and 52 weeks.

Study sample: The study sample will consist of 30 individuals at UHR between 16 and 40 years of age.

Main outcome variable: Changes in the positive subscale score as a measure of positive symptoms of the Positive and Negative Syndrome Scale (PANSS) Secondary outcome variables: (i) Changes in SOFAS score; (ii) Changes in metacognitive biases and beliefs; (iii) Changes in PANSS total score Power analysis: The aim of this pilot study is to better understand the magnitude of the treatment effect and its variability, such that future studies can be properly powered. A sample size of 15 in each group was decided upon, with an asymptotic, two-sided 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

(i) Age 16-40 years; (ii) individuals belonging to either one of the following two groups:

* attenuated psychotic symptoms (APS): Experience of subthreshold, attenuated forms of positive psychotic symptoms including ideas of reference, odd beliefs or magical thinking, perceptual disturbance, paranoid ideation, odd thinking and speech, odd behavior and appearance, at least several times per week within the last year, present for at least one week and no longer than five years, according to the criteria operationalized in the Comprehensive Assessment of At Risk Mental State (CAARMS) interview (Yung et al., 2003);
* brief limited intermittent psychotic symptoms (BLIPS): Episodes of frank psychotic symptoms that have not lasted longer than a week and have spontaneously abated, according to the criteria operationalized in the CAARMS interview (Yung et al., 2003); (iii) ability to give informed consent and to follow study procedures

Exclusion Criteria:

(i) Past history of a treated or untreated manifest psychotic episode of one week's duration or longer (ii) Increases of dosages of antipsychotic medications - if any is given at all - within the last two weeks and/or clinical necessity for dosage increases at time of inclusion; (iii) Past neuroleptic exposure exceeding a total lifetime haloperidol dose of 50 mg (equivalent doses as referred to in Gardner, Murphy, O'Donnell, Centorrino, and Baldessarini (2010)); (iv) Acute suicidality or acute aggressive behavior; (v) Current attenuated symptoms that are entirely explained by acute intoxication (e.g., current attenuated symptoms entirely explained by LSD use) (vi) Organic brain disease (e.g. epilepsy, inflammatory brain disease etc.); (vii) Any other physical illness with psychotropic effect, if not stabilized; (viii) Diagnosis of a serious developmental disorder, e.g. Asperger ́s syndrome; (ix) Premorbid IQ lower than 70; (x) Inadequate knowledge of German language

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change Positive and Negativ Syndrome Scale (PANSS) positive subscale | 12, 26, 52 weeks
  The positive subscale of the PANSS is a scale rating the positive psychotic symptoms of an individual, where higher scores mean more symptoms. It consists of 7 items, where each item is rated from 1-7. So the minimum score is 7 and the maximum score is 49.

SECONDARY OUTCOMES:
Change in the Social and Occupational Functioning Assessment Scale (SOFAS) scores | 12, 26, 52 weeks
  The SOFAS is a scale used to rate current social and occupational functioning of an individual.To be rated a reduction in functioning must be directly related to mental or physical health issues. The scale is rated between 0-100, where higher scores mean higher functioning.
Change in metacognitive biases: Metacognitions-Questionnaire-30 (MCQ-30), Beck Cognitive Insight Scale (BCIS), Fish Task, Davos Assessment of Cognitive Biases Scale (DACOBS), Reading the Mind in the Eyes (RMET) Test. | 12, 26, 52 weeks
  MCQ-30 is a 65-item scale to assess metacognition. Each item is rated on a 4-point scale.
  BCIS is a 15-items self administered scale assessing cognitive insight. It has a rating from 1-4 (do not agree to agree completely). Fish task is used to assess jumping to conclusion; the patient has the task to decide whether a fish comes from pond A or B according to subjective probabilities. RMET is a 36-item test to assess Theory of Mind; one has to guess the correct adjective best describing a set of eyes among 4 adjectives presented; each correct answer is rated with 1 point; a higher score meaning better Theory of mind. DACOBS is a 42 items scale used to assess cognitive biases specific to positive symptoms; each item is rated from 1-7, 7 subscales are calculated from the items, higher scores meaning more cognitive biases.
Change in Positive and Negative Syndrome Scale (PANSS) total scores | 12, 26, 52 weeks
  The PANSS is a scale to rate positive, negative an global symptoms in schizophrenia. The positive subscale consists of 7 items, as well as the negative subscale, the global subscale consists of 16 items. Each item is rated from 1-7, where higher scores mean more severe symptoms. The minimum PANSS total score is 30, the maximum is 210.

CONTACTS AND LOCATIONS:
Overall Officials: Nilufar Mossaheb, MD, Principal Investigator — Medical Univ. Vienna, Clinical Division of Social Psychiatry
Locations (2):
- Austria (2):
  - Department of Child and Adolescent Psychiatry, Vienna
  - Department of Psychiatry and Psychotherapy, Vienna

IPD SHARING:
Plan to Share IPD: No